CLINICAL TRIAL: NCT01390480
Title: Placebo Controlled Pilot Study on Effects of Vitamin D Supplementation in Subjects With New Onset of Type 1 Diabetes on Immunological, Endocrine and Metabolic Parameters: Step 2 in the Austrian Diabetes Prevention Programme
Brief Title: Effects of Vitamin D Supplementation in Subjects With New Onset of Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENM-DA-017
Record Dates: First submitted 2011-05-23; First posted 2011-07-11 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes
Keywords: vitamin D; Autoimmune disease; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Diabetes Mellitus | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): peanut oil
  Interventions: Drug: Cholecalciferol
- Vitamin D (Oleovit®) (Active Comparator): cholecalciferol
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — weekly dose (based on 70 IU/kg bodyweight/day) orally
  Other Names: intervention: Oleovit D3; Placebo: peanut oil

SUMMARY:
In this placebo controlled study the investigators aim to investigate the effects of vitamin D supplementation in subjects with new onset of type 1 diabetes on immunological, endocrine and metabolic parameters.

DETAILED DESCRIPTION:
This is a bicentric, randomized placebo controlled, double blind study, with the aim to evaluate the effect of vitamin D supplementation in subjects with new onset of type 1 diabetes on immunological, endocrine and metabolic parameters.

The primary study goal is to evaluate the influence of vitamin D supplementation on the number and function of the master regulatory T-cells under controlled conditions within 13 months. The secondary study goals are a comprehensive immune phenotyping to determine whether Vit D produces changes consistent with a general improvement in immune homeostasis that supports ß-cell tolerating interventions, the assessment of ß-cell function in all subjects to obtain preliminary data on the effects of Vit D on ß-cell survival.

ELIGIBILITY:
Inclusion Criteria:

* males or females > 6 years
* new onset of type 1 diabetes (3 months)

Exclusion Criteria:

* pregnancy
* hypercalcemia (>2,65 mmol/L)
* chronic disease including a long-term medication over 4 weeks per year (except type 1 diabetes)

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Increase and function of regulatory T-cells | 13 months
  The level and function of the regulatory T-cells will be compared between the two groups.

SECONDARY OUTCOMES:
Immunophenotyping | 13 months
  The effect of vitamin D on circulating immune cells and cytokine secretion at basal, after 3, 6 and 12 months.
Insulin secretion | 13 months
  Insulin secretion assessed with a mixed meal tolerance test will be performed basal, after 3, 6 and 12 months.
Calcium levels | 13 months
  Serum calcium levels will be measured basal, after 1,3,6,9 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria

REFERENCES:
- [Derived] Treiber G, Prietl B, Frohlich-Reiterer E, Lechner E, Ribitsch A, Fritsch M, Rami-Merhar B, Steigleder-Schweiger C, Graninger W, Borkenstein M, Pieber TR. Cholecalciferol supplementation improves suppressive capacity of regulatory T-cells in young patients with new-onset type 1 diabetes mellitus - A randomized clinical trial. Clin Immunol. 2015 Dec;161(2):217-24. doi: 10.1016/j.clim.2015.08.002. Epub 2015 Aug 12. PMID 26277548